CLINICAL TRIAL: NCT03066921
Title: Evaluation of the Effects of a Probiotic Formulation in Hemodialysis Patients
Brief Title: Evaluation Of The Efficacy of a Strain-Specific Probiotic Formulation in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paik Seong Lim (Other)
Responsible Party: Sponsor-Investigator, Paik Seong Lim, National Science Council, Tungs' Taichung Metroharbour Hospital
Organization: Tungs' Taichung Metroharbour Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 104012
Record Dates: First submitted 2017-02-20; First posted 2017-03-01 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: End Stage Renal Disease
Keywords: Lactic acid bacteria; dyslipidemia uremic toxins; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Randomized placebo controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo packet will be given at a dose of one sachet thrice daily for 24 weeks; Placebo packet contain all excipients as present in packets (without the 3 strains of bacteria as mentioned above).
  Interventions: Dietary Supplement: Placebo
- Probiotic packet (Experimental): Probiotic formulation will be given at a dose of one packet thrice daily for 24 weeks, amounting to a total of 300 billion colony forming units(CFU)/day. Each packet contains 100 billion viable lyophilized bacteria of three strains of Lactobacillus viz Lactococcus lactis subsp. Lactis LL358 (BCRC910699)、Lactobacillus salivarius LS159 (BCRC910700) and Lactobacillus pentosus and excipients.
  Interventions: Dietary Supplement: Probiotic packet

INTERVENTIONS:
Dietary Supplement: Probiotic packet — Probiotic formulation will be given at a dose of one packet thrice daily for 24 weeks, amounting to a total of 300 billion colony forming units(CFU)/day. Each packet contains 100 billion viable lyophilized bacteria of three strains of Lactobacillus viz Lactococcus lactis subsp. Lactis LL358 (BCRC910699)、Lactobacillus salivarius LS159 (BCRC910700) and Lactobacillus pentosus and excipients.
  Arms: Probiotic packet
Dietary Supplement: Placebo — Placebo packet will be given at a dose of one sachet thrice daily for 24 weeks; Placebo packet contain all excipients as present in packets (without the 3 strains of bacteria as mentioned above).
  Arms: Placebo

SUMMARY:
Previous studies found that lactic acid bacteria could inhibit the activity of the performance of aristolochic acids (AAs) and improve apoptosis of proximal tubular epithelial cells (NRK-52E) and renal fibrosis on rats. The aim of this study is to assessment a novel health food of lactic acid bacteria for preventing renal dysfunction and replacing or assisting conventional drug treatment. This study in 300 hemodialysis patients with dialysis quality assessment index (KT/V, urea reduction ratio (URR), albumin, prealbumin, Hb, CRP…) screened for more than three months, and the stability of the situation in dialysis patients. They will be divided into two groups in order to conduct ergonomic assessments. One group maintains their original diet and medicine. The other group will take the novel lactic acid bacteria and placebo (1x1011 cfu/3±0.2 g/bag) in every morning and evening after their meals. The effect of 0, 6, 12, 18, 24 weeks of the novel lactic acid bacteria will be assessed after starvation for 4 weeks. Group C was the control group did not give any test samples, but continued to observe. The overall goal of the aforementioned study is to develop a novel food product of lactic acid bacteria which can improve dialysis quality for hemodialysis patients. The investigators hope that this novel product can get a patent and be commercialized.

DETAILED DESCRIPTION:
Background:

Insulin resistance (IR) and its associated metabolic disorders are common features of chronic kidney disease (CKD)and accumulating evidence suggested they are important contributors for the cardiovascular burden of CKD patients. In recent years, the modification of the intestinal ﬂora and activation of inflammation pathways have been implicated in the pathogenesis of IR in patients suffering from metabolic syndrome. These important discoveries have led to major advances in understanding the mechanisms of uraemia-induced IR. Furthermore, recent studies show impairment of the intestinal barrier and renal function function as well as changes in the composition of the gut microbiome can contribute to the prevailing inflammation, and gut-derived uremic toxins. Some of these uraemic toxins have been linked to the pathogenesis of IR.

Probiotics is one of the functional foods believed to mediate their health promoting activities through modulating the composition of the gut health. Ingestion of probiotics has been shown not only to influence gut microbiota composition but also the secretion of the gut hormones that ameliorate insulin resistance in animal models. Limited trials in human also showed that supplementation with probiotic not only affect glucose homeostasis, but improved other diabetes related comorbidities such as metabolic syndrome, hypertension, and hyperlipidemia. It also increasing clear that many of the multifactorial physiological functions of gut bacteria are highly strain specific, preselection of appropriate probiotic strains based on their expression of functional biomarkers is critical

Objectives and hypotheses:

To address this research gap, this randomized controlled trial is proposed to determine the efficacy of probiotic formulation to improve metabolic profile and reduction of uremic toxins through modulating gut microbiota composition and gut immune function in hemodialysis patients.The investigators hypothesized that the probiotic supplementations will improve blood glucose control as well as other related metabolic aberrations and lower the levels of gut-derived uremic toxins.

Methodology:

This is a single center, double blind randomized parallel group control trial with 6 months probiotic formulation with strain specific lactobacillus or placebo. After screening the eligible subjects will be selected. Then, after consent taking and 4 weeks of washout period, participants will be randomly assigned to either receive probiotic formulation or placebo for 6 months. Measurements of blood parameters including glycemic control related parameters, lipid profile, nutritional markers, inflammatory markers and uremic toxins. Nutritional assessments, quality of life assessment and anthropometry measurements will take place at baseline, and after 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Both sexes aged between 20-75 years.
2. Received stable hemodialysis at least 3 months.
3. Written informed consent.

Exclusion Criteria:

1. patients with severe infections, severe heart disease and liver disease, malignancy, autoimmune disorders, severe malnutrition, or clinical conditions requiring oral nutrition supplements;
2. Inability to follow protocol.
3. patients with known gastro-intestinal disease (i.e.,inflammatory bowel disease,crohn's disease,ulcerative colitis)
4. Use of antibiotics, prebiotics or probiotics and immunosuppression medications in the past 4 weeks
5. Pregnancy or wishing/trying to get pregnant

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Triglyceride/HDL cholesterol ratio at 3 months, 6 months and 3 months after the trial | baseline,3 months, 6 months and 3 months after the trial
  Plasma triglycerides are measured by enzymatic methods. High-density lipoprotein (HDL) cholesterol is measured in the supernatant after sodium phosphotungstate/magnesium chloride precipitation.

SECONDARY OUTCOMES:
Plasma concentrations of typical gut-derived uremic toxins(Indoxyl sulfate and p-cresyl sulfate) | baseline,3 months, 6 months and 3 months after the trial
  All uremic toxins are measured by a high performance liquid chromatography method and fluorescence detection method.
plasma concentrations of inflammatory biomarkers | baseline,3 months, 6 months and 3 months after the trial
  Interleukin-6 (IL-6) level is measured by an immunoenzymatic method, and C reactive protein (CRP) levels is measured by an immunonephelometric method.
plasma concentrations of microbial translocation biomarkers | baseline,3 months, 6 months and 3 months after the trial
  LBP and sCD14 are measured using an enzyme-linked immunosorbent assay (ELISA).
Quality of life | baseline and 6 months
  Assessed with the Medical Outcomes Study Short Form 36-Item Health Survey (SF-36)
Nutritional Status | baseline and 6 months
  Assessment with Subjective Global Assesment(SGA) and Mini Nutritional Assessment (MNA)
Gut function questionnaire as a measure of tolerability | Symptoms during first month
  Questionnaire is used to assess the tolerability of the probiotic supplementation. Questionnaire includes questions on frequency and severity of flatulence and bloating, occurrence of diarrhea, frequency of defecation, and texture of feces using a stool chart.

CONTACTS AND LOCATIONS:
Overall Officials: Paik Seong Lim, PhD, Principal Investigator — Tungs' Taichung Metroharbour Hospital
Locations (1):
- Tungs' Taichung MetroHarbour Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lim PS, Wang HF, Lee MC, Chiu LS, Wu MY, Chang WC, Wu TK. The Efficacy of Lactobacillus-Containing Probiotic Supplementation in Hemodialysis Patients: A Randomized, Double-Blind, Placebo-Controlled Trial. J Ren Nutr. 2021 Mar;31(2):189-198. doi: 10.1053/j.jrn.2020.07.002. Epub 2020 Sep 6. PMID 32900583